CLINICAL TRIAL: NCT06757959
Title: Effectiveness of Wet Needling Technique in Patients of Patellofemoral Pain Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/756
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group I (Experimental)
  Interventions: Combination Product: Wet Needling
- Interventional group II (Active Comparator)
  Interventions: Diagnostic Test: Kinesiotaping

INTERVENTIONS:
Combination Product: Wet Needling — This involve the use of needles to inject a local anesthetics into trigger points or areas of muscle tightness around the knee particularly in the quadriceps surrounding soft tissue implicated in patellofemoral pain syndrome .To reduce localized pain, release muscle tension and improve tissue function.
  Arms: Interventional group I
Diagnostic Test: Kinesiotaping — Application of kinesiotape around knee joint or quadricep following a specific technique aimed at reducing pain and improving joint stability . The tape is typically applied to encourge proper movement patterns , reducing swelling and provide sensory feedback to brain. Strengthening exercises : To strenghthen the quadriceps , gluteal muscles and other key stabilizing muscles of lower limbs. This is aimed at reducing the mechanical stress on the joint and improve overall function.
  Arms: Interventional group II

SUMMARY:
This study evaluate the effectiveness of wet needling technique in reducing pain, improving function and enhancing the quality of life in patellofemoral pain syndrome patient.Patellofemoral pain syndrome is a common knee condition that significantly affects physical activity and quality of life .

DETAILED DESCRIPTION:
This study aims to determine wether integrating wet needling into a kinesiotaping and strenghthening exercises regimen provides enhanced outcomes for patellofemoral pain syndrome patients .Wet needling combined with kinesiotaping and strengthening eexercises provides superior pain relief and functional improvement .Participant will divided into two groups : one will recieve treatment using wet needling with kinesiotaping and strengthening exercises , and the other recieve kinesiotaping and strengthening exercises.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20-35
* unilateral , prepatellar or retropatellar pain unrelated to trauma for atleast 3 month , agerevated witrh atleast 2 daily activities such as prolonged sitting, squatting , kneeling , running or stairs climbing.
* Positive clarkes sign.
* Average pain in the previous week >3 on numeric pain rating scale. Kujala questionnaire score <85of 100.
* Active trigger points in gluets and quadriceps.
* Presence of palpable taut band in muscle and typical reffered pain .

Exclusion Criteria:

* Bilateral anterior knee pain.
* Patients with fracture of knee joint , dislocation of patella , previous knee or ankle surgery and ligament or meniscus injury .
* Marked structural deformity and known pathological condition of back , hip and ankle . Any metabolic or neurological disease such as diabetes or radicular pain . Physical therapy for knee pain within the previous year .

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Numeric rating pain scale (NRPS ) | 12 Months
  Numeric rating pain scale (NRPS ) is utilized as the primmary outcome measure to quantifying the intenstiy of pain. It consists of 0 to 10 scale , where the pain rates on the based of intensity .
Kujala score | 12 Months
  It is used to asses the severity of symptoms and functional limitation in individuals with patellofemoral pain syndrome . It focuses on pain , functional limitations and impact of the condition on daily activities. The kujala score consist of 13items . Each question is scored from 0 to 5 based on the severity of symptoms . The total score is the sum of all 13 items , with apossible range from 0 to 100 . 100 indicate no symptooms and normal function.0 indicates symptoms and total disability . <65:severe PFPS , with significant pain and functional restrictions .65-84 : Moderate PFPS, with noticeable pain and some functional limmitations. 85-100: Mild PFPS or recovery, with minimal symptoms and good function.

CONTACTS AND LOCATIONS:
Locations (1):
- Medsol medical solutions sahiwal, Street between qureshi and total pump , mall mandi chowk, Sahiwal, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No